CLINICAL TRIAL: NCT05522088
Title: Effectiveness of Prophylactic Bolus Ephedrine Versus Norepinephrine for Management of Post Spinal Hypotension During Elective Caesarean Section in Resource Limited Setting: a Prospective Cohort Study
Brief Title: Effectiveness of Prophylactic Bolus Ephedrine Versus Norepinephrine for Management of Post Spinal Hypotension
Status: Completed | Type: Observational
Sponsor: Wachemo University (Other)
Responsible Party: Principal Investigator, Mitiku Desalegn, Mr, Wachemo University
Other Study IDs: NE2323
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Comparing Ephedrine With Norepinephrine for Mangement Postspinal Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study was conducted to compare the effectiveness of ephedrine versus norepinephrine for management of hypotension after spinal anesthesia for mothers undergoing elective cesarean section

ELIGIBILITY:
Inclusion Criteria:

* ASA class II and ages ranging from 18-35 years were included in the study

Exclusion Criteria:

* pregnant women with preeclampsia/eclampsia, baseline hypertension (SBP> 140 mm Hg), BMI> 30 kg/m2, failed spinal, spinal anaesthesia converted to general anaesthesia, contraindication for spinal anaesthesia and mother with cardiovascular, renal or hepatic disease.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: All pregnant women undergoing elective cesarean section fulfills the inclusion criteria were the source population
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
to compare mean blood pressure (MAP) between the groups | From March,01 to April, 30/2022

CONTACTS AND LOCATIONS:
Locations (1):
- Wachemo University, Hosa’ina, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Desalegn M, Shitemaw T, Tamrat H. Effectiveness of Prophylactic Bolus Ephedrine Versus Norepinephrine for Management of Postspinal Hypotension during Elective Caesarean Section in Resource Limited Setting: A Prospective Cohort Study. Anesthesiol Res Pract. 2022 Oct 3;2022:7170301. doi: 10.1155/2022/7170301. eCollection 2022. PMID 36225250